CLINICAL TRIAL: NCT00116636
Title: A Phase II, Open Label, Single Arm Study of the 48-Week Virologic and Immunologic Response to Lopinavir/Ritonavir (Kaletra) as a Single Agent in a Cohort of HIV Positive Adult Patients
Brief Title: Study of the 48-Week Virologic and Immunologic Response to Lopinavir/Ritonavir (Kaletra) in HIV Positive Adult Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutic Concepts (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 70-1002-064
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2005-06

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination

INTERVENTIONS:
Drug: Kaletra

SUMMARY:
Expected Enrollment: 40 patients

Study Start Date: June 2005

Study Objectives:

* To conduct a pilot study to assess the safety, tolerability, and antiviral activity of Kaletra 400/100 mg taken twice a day (bid) in antiretroviral (ARV)-naïve HIV-infected patients at Week 48

Primary Objectives:

* To determine the proportion of patients with HIV RNA <400 copies/mL at weeks 24 and 48
* To determine the proportion of patients with HIV RNA < 50 at weeks 24 and 48
* To elucidate the specific adverse event (AE) profile of Kaletra single agent therapy

Secondary Objectives:

* To assess the proportion of patients below the limit of quantification (LOQ) at each visit. Patients will be observed at baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48.
* To determine the time to HIV RNA reaching <400 and <50 copies/mL
* To determine the time to virologic failure
* To assess change from baseline at each visit for HIV RNA and CD4 count at weeks 4, 8, 12, 24 and 48.
* To assess changes in genotype from baseline to time of confirmed virologic failure (2 consecutive HIV RNA measurements >400 copies/mL after suppressing to <400 copies/mL) or at time of treatment intensification.
* To characterize changes in lipid and triglyceride concentrations over time and the effect of treatment with appropriate drugs (fibrate or statin, if necessary) on these elevations.
* To evaluate the safety and tolerability of subjects through 48 weeks of drug exposure.
* To describe virologic response following intensification in Kaletra single agent virologic failures

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 RNA ≥ 2000 copies/mL by Roche Amplicor 1.5v Primer
* CD4 count -< 400
* CD4 count > 400, with documented understanding of DHHS recommendations related to risks and benefits of early treatment initiation, and stated desire for treatment based upon one of the following conditions: (reference: DHHS guidelines) *Viral load > 100,000 copies; *Symptomatic HIV infection other than an active opportunistic infection - CDC Category B or C condition; *Desire for potential immune function preservation; *Desire for potential decreased risk of HIV transmission to uninfected partner; *Desire for potential prolongation of disease-free survival
* ≥ 18 years of age
* Cognitive ability to understand and provide written informed consent and willingness to participate in and comply with the study protocol
* PI -naïve or has < 7 days of prior ART with any licensed or investigational compound (NOTE: patients must have no prior PI experience)
* Patient does not currently have or has not been treated for an active opportunistic infection (OI) consistent with CDC definition within 30 days of screening
* Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness
* A female is eligible to enter and participate in this study if she is of: (1) Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal) -OR- (2) Child-bearing potential, has a negative serum pregnancy test at screen, and agrees to one of the following: Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for at least 2 weeks after completion or premature discontinuation from the study to account for elimination of the investigational drug. Should a patient decide to become sexually active during the course of the study, she must be counseled and be willing to use one of the birth control methods listed below: *Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide); *Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion); *Sterilization (female patient or male partner of female patient); *Any other methods with published data showing that the lowest expected failure rate for that method is <1% per year.

NOTE: Data are insufficient to exclude a clinically important interaction of LPV/r with drugs, such as hormonal contraceptives, that are highly metabolized by the cytochrome P450 enzyme system. As a result, hormonal contraception is not considered adequate.

Exclusion Criteria:

* Patient with active AIDS-defining opportunistic infection or disease according to the 1993 CDC AIDS surveillance definition (Clinical Category C) that, in the opinion of the investigator, would preclude the patient from participating in the study.
* Patient has an M184V mutation in reverse transcriptase, or mutations at 10, 20, 32, 46, 47, 48, 50, 54, 71, 73, 82, 84, or 90;
* K65R mutation or 2 or more TAMs at baseline
* History of active substance abuse, excluding cannabis, or psychiatric illness that, in the opinion of the investigator, would preclude compliance with protocol, dosing schedule and assessments.
* Patient is either pregnant at time of screening evaluation or breast-feeding.
* Patient, in the opinion of the investigator, is unlikely to be able to complete the 48-week dosing period and protocol evaluations and assessments or adhere to the study drug regimen.
* Patient suffers from a serious medical condition, such as diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction, which in the opinion of the investigator would compromise the safety of the patient
* Patient has malabsorption syndrome or other gastrointestinal dysfunction, which may interfere with drug absorption or render the patient unable to take oral medication.
* Patient is undergoing interferon therapy for HCV or anticipates undergoing therapy during the course of this trial
* HBV coinfection
* Patient has any of the following laboratory results within 30 days prior to the first dose of study medication: *Hemoglobin concentration < 8.0 g/dL; *Absolute neutrophil count < 750 cells/mm3; *Platelet count <50,000 cells/ mm3; *Aminotransferase (AST, ALT) >3 times ULN; *Serum creatinine >1.5 times the Upper Limits of Normal (ULN)
* Patient has required treatment with radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to entry, or has an anticipated need for these agents within the study period.
* Patient requires treatment with immunomodulating agents, such as systemic corticosteroids, interleukins, or interferon's within 4 weeks prior to study entry, or patients who have received an HIV immunotherapeutic vaccine within 3 months prior to entry. Asthmatic patients using inhaled corticosteroids are eligible for enrollment.
* Patient receiving methadone therapy
* Patients requiring foscarnet therapy or therapy with other agents with documented activity against HIV-1 in vitro.
* Patient prescribed/taking astemizole, terfenadine, cisapride, midazolam, triazolam, flecainide, pimozide, propafenone, St. John's Wort, lovastatin, simvastatin, and rifampin or ergot derivatives
* Patient has a history of allergy to any of the study drugs or any excipients therein.
* In addition, patients non-compliant with study medication during 2 - 4 week study periods despite adherence counseling will not be retained in the study due to increased risk for selective pressure and potential development of protease resistance.
* Patient requires inhaled or intranasal fluticasone.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-06; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA <400 copies/mL at Week 24 and 48
Proportion of patients with plasma HIV-1 RNA < 50 copies/mL at Week 48

SECONDARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA <400 copies/mL or <50 copies/mL at each study visit
Proportion of patients with plasma HIV-1 RNA <50 copies/mL at Weeks 24 and 48 Weeks
Number of weeks until HIV RNA <400 copies/mL and <50 copies/mL, respectively
Change from baseline to each study visit in plasma HIV-1 RNA and CD4+ cell count
Time-averaged change from baseline to Weeks 12, 24 and 48 (AUCMB) in plasma HIV-1 RNA and CD4+cell count
Change in HIV genotype and phenotype in patients who either intensify study therapy or experience virologic rebound
HIV genomic sequence in treatment failures
Adverse events and treatment-limiting toxicities at all time points
Baseline and on-therapy assessment of clinical laboratory parameters
Change from baseline over time in clinical laboratory parameters including fasted triglycerides, total cholesterol, direct HDL cholesterol and LDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Gathe, M.D., Principal Investigator — Therapeutic Concepts, P.A.
Locations (1):
- Therapeutic Concepts, P.A., Houston, Texas, United States

REFERENCES:
- [Background] Mocroft A, Vella S, Benfield TL, Chiesi A, Miller V, Gargalianos P, d'Arminio Monforte A, Yust I, Bruun JN, Phillips AN, Lundgren JD. Changing patterns of mortality across Europe in patients infected with HIV-1. EuroSIDA Study Group. Lancet. 1998 Nov 28;352(9142):1725-30. doi: 10.1016/s0140-6736(98)03201-2. PMID 9848347
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Staszewski S, Morales-Ramirez J, Tashima KT, Rachlis A, Skiest D, Stanford J, Stryker R, Johnson P, Labriola DF, Farina D, Manion DJ, Ruiz NM. Efavirenz plus zidovudine and lamivudine, efavirenz plus indinavir, and indinavir plus zidovudine and lamivudine in the treatment of HIV-1 infection in adults. Study 006 Team. N Engl J Med. 1999 Dec 16;341(25):1865-73. doi: 10.1056/NEJM199912163412501. PMID 10601505
- [Background] Kaletra® (lopinavir/ritonavir) capsules-Complete Product Information
- [Background] Information for Clinical Investigators: Lopinavir (Abbott-157378) V 7.0
- [Background] Kempf et al. Seville 2002
- [Background] Stevens, et al. SOKRATES: Prospective Clinical Trials to Investigate the Evolution of Protease Resistance During Lopinavir/r Treatment. 2003. 1st European Drug Resistance Workshop, Luxemburg
- [Background] Allavena et al. Lopinavir/ritonavir-Efavirenz (LPV/r-EFV) NRTI-sparing Regimen (BIKS study): Preliminary Efficacy and Safety Data. 42nd ICAAC, San Diego 2002, #H-169
- [Background] Lauenroth-Mai & Schuler. Nuc-sparing salvage therapy: Immunological and virological response to a combination of indinavir (IDV) and lopinavir/ritonavir (LPV/r) in intensively pretreated HIV-infected patients with multiple NRTI resistance mutations. 6th IWDTHI, Glasgow 2002.
- [Background] Gathe et al. Pilot Study of the Safety and Efficacy of Lopinavir/Ritonavir (LPV/r) as Single Agent Therapy in HIV-1 ARV Naïve Patients. 44th Annual ICAAC, Washington, DC 2004.
- [Background] Pierone et al. Initial clinical experience with Kaletra (LPV/r) single agent therapy in HIV infection. 2002. HIV DART; Poster 076
- [Background] Pierone et al. Genotypic and phenotypic resistance observations among patients with viremia with on lopinavir/ritonavir "monotherapy". 44th Annual ICAAC, Washington, DC 2004.